CLINICAL TRIAL: NCT01249469
Title: Evaluate the Lightening Effect of the Whitening Cosmetic Product BEX-2011 on Solar Lentigines by Harmonic Generation Microscopy
Brief Title: Evaluate the Lightening Effect of the Whitening Cosmetic Product BEX-2011
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: L'Oreal (Industry)
Responsible Party: Laurent GILBERT, Loreal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201003024M; NTUH201003024M (Registry Identifier: NTUH)
Record Dates: First submitted 2010-11-25; First posted 2010-11-29 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2010-04

CONDITIONS: Solar Lentigines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle (Placebo Comparator): Product application: twice a day in the morning and before sleep for 8 weeks; from D1 to D55, but no application on D27 at night/ D28 in the morning and D55 at night/ D56 in the morning before visit. The product is applied on one side of the hand.
  Interventions: Other: skin whitening cosmetic product
- Skin whitening cosmetic product (Experimental): Product application: twice a day in the morning and before sleep for 8 weeks; from D1 to D55, but no application on D27 at night/ D28 in the morning and D55 at night/ D56 in the morning before visit. The product is applied on one side of the hand.
  Interventions: Other: skin whitening cosmetic product

INTERVENTIONS:
Other: skin whitening cosmetic product — Product application: twice a day in the morning and before sleep for 8 weeks; from D1 to D55, but no application on D27 at night/ D28 in the morning and D55 at night/ D56 in the morning before visit. The product is applied on one side of the hand
  Other Names: BEX-2011

SUMMARY:
Background: Solar lentigines are a common dermatologic condition that manifest as circumscribed single or multiple brownish macules usually located on sun-exposed skin such as face, hands or forearms. An effective, safe, daily-use, homecare whitening product may alleviate the cosmetic concerns for the general population. The efficacy and safety of the previous generation BEX-2009 (Blanc Expert Spot Eraser, L'Oreal, France), a whitening cosmetic product containing ellagic acid, salicylic acid, licorice root extract, etc., has been established in Caucasian and Asian populations with facial solar lentigines.

Objective: The purpose of this placebo-controlled, single-center study is 1) to evaluate the efficacy of the new generation whitening cosmetic product BEX-2011 (Ultimate Whitening Spot Eraser, L'Oreal, France) in the improvement of solar lentigines on the dorsum of hands or forearms, and 2) to evaluate the efficacy of BEX-2011 by harmonic generation microscopy to obtain information of the epidermal melanin continuum, compared to other standard tools for melanin measurement.

DETAILED DESCRIPTION:
Method: 40 subjects, who are non-gravid women between 45 to 65 years old and need to have ≥10 solar lentigines on the forearms/hands, will be recruited. One to three flat lesions which are larger than 4 mm and with the same pigmentation intensity on the left or right forearm/hand, respectively, are designated the target lesions. However, all lesions on the randomly selected side will be treated with BEX-2011 twice a day. The opposite site will be treated with vehicle and is served as the control. Evaluation will be performed at week 0, 4 and 8. At each visit, treated and control spots as well as their surrounding spotless skin will be evaluated using Pigmentation Index Scores, VISIA-CR, SIAscope, Dermascore, and harmonic generation microscopy. Evaluation of the efficacy of whitening will be compared to the baseline and to the control area between week 0 and week 8. Safety will be assessed using clinical monitoring and adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

* 40-65 years old Asian women (skin types III to IV)
* With ≥10 solar lentigines on the forearms or dorsum of hands
* With at least one to three lesions ≥4 mm on the left or right forearm/ dorsum of hand, respectively, which are flat and are at the same pigmentation degree according to the color chart.

Exclusion Criteria:

* Having major treatment, including topical hydroquinone or tretinoin, cryotherapy, electrosurgery, trichloroacetic acid application, laser or intense pulsed light, in the 3 months before the beginning of the study
* Past history of allergy to whitening cosmetic products
* Past history of atopic dermatitis
* Habit of going to the tanning salon or frequent sun exposure longer than 4 hours per day

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
the mean reduction of darkness from baseline in target area after treatment | 8 weeks

SECONDARY OUTCOMES:
the difference of darkness between the treated spots and the control spots | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hua Liao, MD, PhD, Principal Investigator — Department of Dermatology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Farris PK. Combination therapy for solar lentigines. J Drugs Dermatol. 2004 Sep-Oct;3(5 Suppl):S23-6. PMID 15552596
- See also: PubMed — http://www.ncbi.nlm.nih.gov/pubmed